CLINICAL TRIAL: NCT05604053
Title: Motivation Effects During Cued Visual Search
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lehigh University (Other)
Responsible Party: Principal Investigator, Nancy Carlisle, Associate Professor of Psychology and Cognitive Science, Lehigh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2R15EY030247-01A1 (NIH)
Record Dates: First submitted 2022-10-19; First posted 2022-11-03 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: attention; visual search

STUDY DESIGN:
Intervention Model Description: All participants receive each level of visual cue type and motivation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-subjects motivation manipulation (Experimental): Low or high motivation
  Interventions: Behavioral: Motivation Manipulation

INTERVENTIONS:
Behavioral: Motivation Manipulation — On some trials, participants have lower motivation and on other trials participants have higher motivation.

SUMMARY:
In this line of research, we are examining whether motivation increases the utilization of target (positive) or distractor (negative) color cues to improve visual attention performance.

DETAILED DESCRIPTION:
When finding a search target, receiving a target cue or distractor cue can increase search efficiency. We are examining whether we can improve people's use of the cues to aid visual search performance if we increase their motivation through reward or time pressure.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal visual acuity, normal color vision

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-09-17 (Estimated); Study Completion 2024-09-17 (Estimated)

PRIMARY OUTCOMES:
Button Press Reaction Time | During Testing (single day)
  Speed to respond correctly to the target- after participant finds the target shape on a computer screen, they press a button to indicate what shape they see
Button Press Accuracy | During Testing (single day)
  Accuracy of responses to target item- we will measure whether the participants presses the correct button which corresponds to the target shape presented on the computer screen or the incorrect button

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Carlisle, Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymized subject data on Open Science Framework.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication.
Access Criteria: Open Science Framework internet access.